CLINICAL TRIAL: NCT00995449
Title: A Phase 2, Randomized, Placebo-Controlled, Dose-Ranging Study to Evaluate the Safety and Efficacy of the Anti-GM-CSF Monoclonal Antibody KB003 in Subjects With Active Rheumatoid Arthritis and Inadequate Prior Treatment Outcome From Biologic Therapy
Brief Title: Study of KB003 In Biologics-Inadequate Rheumatoid Arthritis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Program refocus
Sponsor: Humanigen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KB003-02
Record Dates: First submitted 2009-10-05; First posted 2009-10-15 (Estimated); Results first posted 2012-09-25 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; Biologics-Inadequate; KB003; GM-CSF
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — lenzilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- KB003 70 mg (Experimental)
  Interventions: Biological: KB003
- KB003 200 mg (Experimental)
  Interventions: Biological: KB003
- KB003 600 mg (Experimental)
  Interventions: Biological: KB003
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo Comparator

INTERVENTIONS:
Biological: KB003 — KB003 IV x5 doses
  Other Names: Recombinant anti-GM-CSF IgG1K monoclonal antibody
  Arms: KB003 200 mg; KB003 600 mg; KB003 70 mg
Other: Placebo Comparator — Placebo IV x5 doses
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, pharmacokinetics (PK), and efficacy of various repeat-dose regimens of KB003 in subjects with active Rheumatoid Arthritis (RA) who have had an inadequate prior treatment outcome from biologic therapy.

ELIGIBILITY:
Inclusion Criteria:

* At least 6 swollen and at least 6 tender joints
* C-reactive Protein (CRP) > Upper Limit Normal (ULN)
* Prior inadequate response from biologic therapy
* Stable regimens of concomitant RA therapies

Exclusion Criteria:

* Unstable medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nestor A. Molfino, MD, MSC, Study Chair — Humanigen, Inc.
Locations (10):
- United States (10):
  - Stanford, California
  - Westlake Village, California
  - Miami, Florida
  - Honolulu, Hawaii
  - Frederick, Maryland
  - Wheaton, Maryland
  - St Louis, Missouri
  - Wilmington, North Carolina
  - Tulsa, Oklahoma
  - Oak Creek, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a two-part study with a safety run-in. The primary objective of the main portion of the study was to evaluate the safety, PK, and efficacy of selected repeat-dose regimens of KB003 in subjects with active moderate to severe rheumatoid arthritis who had an inadequate treatment outcome from prior biologic therapy.
Pre-assignment Details: The safety run-in portion was conducted in a small cohort of 7 active and 2 placebo subjects to evaluate the acceptability of repeat-dose safety. KB003 was administered by intravenous (IV) infusion as a 600 mg dose at wks 0, 2, 4, 8, and 12, with primary safety being evaluated at wk 14 and a follow-up (end of study) safety assessment at wk 30.
Groups:
- KB003 70mg; KB003 200 mg: Dose group not evaluated in this portion of study
- KB003 600 mg: 600 mg, KB003 a monoclonal antibody
- Placebo: Placebo comparator
Period: Overall Study
Arm/Group | KB003 70mg | KB003 200 mg | KB003 600 mg | Placebo
Started | 0 | 0 | 7 | 2
Completed | 0 | 0 | 5 | 2
Not Completed | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | KB003 70mg | KB003 200 mg | KB003 600 mg | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 7 | 2 | 9
Age, Categorical [Number; unit: participants]
  <=18 years |  |  | 0 | 0 | 0
  Between 18 and 65 years |  |  | 5 | 2 | 7
  >=65 years |  |  | 2 | 0 | 2
Gender [Number; unit: participants]
  Female |  |  | 4 | 1 | 5
  Male |  |  | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States |  |  | 7 | 2 | 9

OUTCOME MEASURES:

1. Primary Outcome: This Study Was Initiated With a Safety run-in Period to Evaluate Acceptability of Repeat-dose Safety.
Description: KB003 was administered by intravenous (IV) infusion as a 600 mg dose at weeks 0, 2, 4, 8, and 12, with primary safety being evaluated at week 14 and a follow-up (end of study) safety assessment at week 30. Safety was evaluated by number of participants with treatment-emergent (TE) adverse events (AEs). (TE is defined as ocurring during the 14 week treatment and week 30 follow-up periods)
Time Frame: Weeks 14 & 30
Population: This safety run-in portion of the study was conducted in a small cohort of 7 active (600 mg) and 2 placebo subjects.
Measure: Number; unit: Participants
Arm/Group | KB003 600 mg | Placebo
Number analyzed (Participants) | 7 | 2
Participants | 7 | 2

ADVERSE EVENTS:
Time Frame: Primary safety data was collected at week 14 and a follow-up(end of study) safety assessment at week 30.
Arm/Group | KB003 70mg | KB003 200 mg | KB003 600 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 1/7 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 7/7 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | KB003 70mg (N=0) | KB003 200 mg (N=0) | KB003 600 mg (N=7) | Placebo (N=2)
Abdominal Hernia Obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0/0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | KB003 70mg (N=0) | KB003 200 mg (N=0) | KB003 600 mg (N=7) | Placebo (N=2)
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
Infections and Infestations (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 1 (1)
Muscoskeletal and Connective Tissue Disorders (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nervous System Disorders (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Psychiatric Disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Cardiac Disorders (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury, Poisoning and Procedural Complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vascular Disorders (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated upon completion of safety run-in due to program refocus.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor has right of first publication of trial results, which will be a joint, multi-center publication of the study results from all appropriate sites contributing data, analysis and comments.